CLINICAL TRIAL: NCT06953869
Title: A Multicenter, Double-Blind, Randomized Study to Evaluate the Effects of Tasimelteon vs. Placebo in Treating Pediatric Insomnia
Brief Title: Evaluating the Effects of Tasimelteon vs. Placebo in Treating Pediatric Insomnia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VEC-162-3108
Record Dates: First submitted 2025-04-01; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-01

CONDITIONS: Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tasimelteon (Experimental)
  Interventions: Drug: Tasimelteon Oral Suspension
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tasimelteon Oral Suspension — Single daily dose, weight-based liquid suspension formulation.
  Arms: Tasimelteon
Drug: Placebo — Placebo comparator.
  Arms: Placebo

SUMMARY:
This is a multicenter, double-blind, randomized study to evaluate the efficacy and safety of a daily single oral dose of tasimelteon and matching placebo in male and female pediatric participants with insomnia disorder.

ELIGIBILITY:
Inclusion Criteria:

* Ability and acceptance to provide written informed consent of the participant or legal guardian (and assent as required).
* Confirmed clinical diagnosis of insomnia disorder
* Males and Females between 2 and 17 years, inclusive.
* The sleep disturbance must not be a result of another medication.

Exclusion Criteria:

* Inability to dose daily with tasimelteon or previous intolerance to tasimelteon.
* Indication of impaired liver function.
* Pregnant or lactating females.
* A positive test for drugs of abuse.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 420 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in sleep latency, as measured by daily sleep diary. | 12 Weeks

SECONDARY OUTCOMES:
Change in nighttime subjective sleep parameters, such as sleep quality, as measured by sleep diary. | 12 Weeks
Change in nighttime subjective sleep parameters, such as sleep time, as measured by sleep diary. | 12 Weeks
Change in daytime functioning, as measured by questionnaire. | 12 Weeks
Change in behavior, as measured by questionnaire. | 12 Weeks
Change in nighttime objective sleep parameters such as sleep time, as measured by actigraphy. | 12 Weeks
Assessment of safety and tolerability of daily single dose of tasimelteon, as measured by spontaneous reporting of adverse events (AEs). | 12 Weeks

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Vanda Investigational Site, Winter Park, Florida
  - Vanda Investigational Site, Charlotte, North Carolina
  - Vanda Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No